CLINICAL TRIAL: NCT05914818
Title: Proof of Concept of Pediatric and Adolescent EXPLORER V2 Exoskeleton in Children With Neurological and Neuromuscular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MarsiBionics (Industry)
Collaborators: National Research Council, Spain (Other Government); Hospital Infantil Universitario Niño Jesús, Madrid, Spain (Other); Hospital Universitario La Paz (Other); Hospital Universitario 12 de Octubre (Other); Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EXP-P-VAL
Record Dates: First submitted 2023-05-30; First posted 2023-06-22 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-08

CONDITIONS: Cerebral Palsy; Acquired Brain Injury; Neuromuscular Diseases in Children
Keywords: exoskeleton; cerebral palsy; acquired brain injury; neuromuscular disease; gait; rehabilitation
MeSH Terms: conditions — Cerebral Palsy; Brain Injuries; Neuromuscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EXPLORER V2 (Experimental): 1 session with the exoskeleton EXPLORER V2 in healthy subjects 3 sessions with the exoskeleton EXPLORER V2 in subjects with disease
  Interventions: Device: EXPLORER V2

INTERVENTIONS:
Device: EXPLORER V2 — 4 sessions of use of the exoskeleton, 1 in a laboratory of gait analysis and 3 in the home and the community of the participants

SUMMARY:
The goal of this clinical trial is to analyze the usability and safety of the prototype gait exoskeleton EXPLORE V2 in children with neurological and neuromuscular disease.

Participants will use the exoskeletons in their home and the community and variables regarding safety and usability will be measured and recorded.

DETAILED DESCRIPTION:
Neurological and neuromuscular diseases are the main cause of motor disability in children, leading to the inability to stand and walk in many cases. Exoskeletons are a useful tool in the rehabilitation of these children, but most of them are designed to be used in the clinical setting. EXPLORER V2 is a prototype of a robotic gait exoskeleton designed to assist gait in children with motor disability in their homes and the community. The aim of this study is to analyze the safety and usability of the EXPLORER V2 as a proof of concept.

A test phase will be conducted in healthy volunteers (phase 0) as a proof of concept with the aim of evaluating safety and usability in healthy participants prior to the use of the device in children with neurological and neuromuscular disease (phases 1 and 2). After this, participants will use the exoskeleton in 4 different ocassions, 1 in a laboratory of gait analysis and 3 in their homes and the community.

ELIGIBILITY:
Inclusion Criteria:

* Medical authorization for standing, gait training and weight bearing.
* Informed consent signed by legal guardians.
* Maximum user weight of 35 kg.
* Hip width (between greater trochanteres) ≤40 cm.
* Length of the thigh (distance from the greater trochanter to the lateral condyle of the tibia) from 21cm to 36cm.
* Tibia leg length (distance from the lateral condyle of the tibia to the lateral malleolus) from 20cm to 35cm.
* Shoe size ≤38 (EU)

Exclusion Criteria:

* Spasticity equal to 4 on the Modified Ashworth Scale at the time of use of the device.
* More than 20º of hip and/or knee flessum at the time of using the exoskeleton.
* Necessity to walk with 15 of hip abduction.
* Skin lesion on parts of the lower extremities that are in contact with the device.
* Scheduled surgery scheduled during the study period.
* History of fracture without trauma. History of bone fracture traumatic in lower extremities or pelvic girdle in the last 3 months.
* Presence of other conditions causing exercise intolerance (such as uncontrolled hypertension, coronary artery disease, arrhythmia, congestive heart failure, severe pulmonary disease).
* Conductual disorders that may interfere with the use of the device or their participation in the study, like impulsiveness or the inability to understand simple comands.
* Allergy to any of the EXPLORER materials: cotton, nylon, polyester, PPS, PEEK or ABS.

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-06-23 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Serious Adverse Events | through study completion, along 6 weeks
  occurrence of any serious adverse event to the participant or the caregiver
Falls prevalence | through study completion, along 6 weeks
  Number of falling events ocurred from the participant or caregiver
Skin integrity | through study completion, along 6 weeks
  Ocurrence of any injury of the skin in the areas of contact and produced by the use of the exoskeleton
Pain (Visual Analogic Scale) | through study completion, along 6 weeks
  pain measured by the Visual Analogic Scale (VAS) by the participant and the caregiver
Spasticity | through study completion, along 6 weeks
  spasticity measured by the Modified Ashworth Scale (MAS)
Kinematic data during gait | Once, during the first session with the exoskeleton
  Kinematic values for each joint of the lower limb during gait, assessed by photogrammetry in a gait analysis laboratory both in healthy subjects and participants with disease
Donning and doffing time | through study completion, along 6 weeks
  Time to don and doff the device to each participant
Heart rate | through study completion, along 6 weeks
  measurement of heart rate when medical prescription
Blood pressure | through study completion, along 6 weeks
  measurement of blood pressure when medical prescription
Oxygen saturation | through study completion, along 6 weeks
  measurement of Oxygen saturation when medical prescription
Participant satisfaction | at the end of the intervention, 6th week
  Satisfaction of the participant (caregiver) with the devicem measured by the Quebec User Evaluation of Satisfaction with Assistive Technology 2.0.
Number of steps | through study completion, along 6 weeks
  Number of steps taken with the exoskeleton provided by the device
Walking time | through study completion, along 6 weeks
  Walking time while using the exoskeleton provided by the device
Interventions of the investigators | through study completion, along 6 weeks
  The amount of times that the investigators have to intervene in the session in order to avoid damage when the device is being used by the caregiver

SECONDARY OUTCOMES:
Acceptability | At the end of the study, 6th week
  Analysis of the drop-out rate during the study period
Accesssibility of the participant | through study completion, along 6 weeks
  Rate of the participants suitable to use the device
Accesssibility of the house | through study completion, along 6 weeks
  Rate of the houses suitable to use the device
Accesssibility of the exterior spaces | through study completion, along 6 weeks
  Rate of the exterior spaces that are suitable to use the device

CONTACTS AND LOCATIONS:
Overall Officials: Olga Arroyo Riaño, Principal Investigator — Hospital Universitario Gregorio Marañón; María Teresa Vara Arias, Principal Investigator — Hospital Infantil Universitario Niño Jesús; Ignacio Martínez Caballero, Principal Investigator — Hospital Infantil Universitario Niño Jesús; Sandra Espinosa García, Principal Investigator — Hospital Univsersitario La Paz; Sofía García de las Peñas, Principal Investigator — Hospital 12 de Octubre; Elena García Armada, Principal Investigator — National Research Council, Spain; Eva Barquín Santos, Principal Investigator — Marsi Bionics S L
Locations (5):
- Spain (5):
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Infantil Universitario Niño Jesús-Servicio de Rehabilitación, Madrid
  - Hospital Universitario Niño Jesús-Servicio de Neuro Ortopedia, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid